CLINICAL TRIAL: NCT06484062
Title: A Phase I Study Evaluating the Safety of Cirtuvivint as Monotherapy and in Combination With ASTX727 in Patients With Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML)
Brief Title: Testing the Anti-cancer Drug, Cirtuvivint, and Its Combination With ASTX727 to Improve Outcomes in Patients With Acute Myeloid Leukemia and Myelodysplastic Syndromes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-05326; NCI-2024-05326 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10674 (Other: Dana-Farber - Harvard Cancer Center LAO); 10674 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2024-06-29; First posted 2024-07-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Myelodysplastic Syndrome/Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Recurrent Myelodysplastic Syndrome/Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome; Refractory Myelodysplastic Syndrome/Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; GATA2 Deficiency | interventions — Specimen Handling; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort I (cirtuvivint) (Experimental): Patients receive cirtuvivint PO QD on days 1-5, 8-12, 15-19, and 22-26 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA at screening. In addition, patients undergo blood sample collection and bone marrow aspiration at screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cirtuvivint; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan
- Cohort II (cirtuvivint) (Experimental): Patients receive cirtuvivint PO QD on days 1, 4, 8, 11, 15, 18, 22, and 25 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA at screening. In addition, patients undergo blood sample collection and bone marrow aspiration at screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cirtuvivint; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan
- Cohort III (cirtuvivint, ASTX727) (Experimental): Patients receive cirtuvivint PO QD on days 1, 4, 8, 11, 15, 18, 22, and 25 and ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA at screening. In addition, patients undergo blood sample collection and bone marrow aspiration at screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cirtuvivint; Drug: Decitabine and Cedazuridine; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Drug: Cirtuvivint — Given PO
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
  Arms: Cohort III (cirtuvivint, ASTX727)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of SM08502 (cirtuvivint) alone and in combination with ASTX727 in treating patients with acute myeloid leukemia (AML) and myelodysplastic syndromes (MDS). Cirtuvivint may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. ASTX727 is a combination of two drugs, decitabine and cedazuridine. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Giving cirtuvivint alone or in combination with ASTX727 may be safe, tolerable, and/or effective in treating patients with AML and MDS.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase 2 dose (RP2D) of SM08502 (cirtuvivint) as monotherapy in relapsed/refractory (R/R) acute myeloid leukemia (AML) and myelodysplastic syndromes (MDS) (Cohort I and II) and in combination with decitabine and cedazuridine (ASTX727) in frontline MDS (Cohort III).

SECONDARY OBJECTIVES:

I. To assess the safety/tolerability of SM08502 (cirtuvivint) as monotherapy in R/R AML and MDS (Cohort I and II) and in combination with ASTX727 in frontline MDS (Cohort III).

II. To assess the pharmacokinetics (PK), and pharmacodynamics (PD) of SM08502 (cirtuvivint) as monotherapy in R/R AML and MDS (Cohort I and II) and in combination with ASTX727 in frontline MDS (Cohort III).

III. To determine the preliminary efficacy of the combination of SM08502 (cirtuvivint) as monotherapy in R/R AML and MDS (Cohort I and II) and in combination with ASTX727 in frontline MDS (Cohort III) by assessing the response rate as defined by the 2022 European LeukemiaNet (ELN) response criteria for AML (Döhner et al., 2022) and International Working Group (IWG) 2023 response criteria for MDS (Zeidan et al., 2023).

IV. To explore survival outcomes achieved with SM08502 (cirtuvivint) as monotherapy in R/R AML and MDS (Cohort I and II) and in combination with ASTX727 in frontline MDS (Cohort III) by assessing 1 year event free survival (EFS) and overall survival (OS) rate.

V. To observe and record anti-tumor activity. VI. To evaluate the best schedule to move forward with in Phase 2.

OUTLINE: This is a dose-escalation study of cirtuvivint as monotherapy. Patients are assigned to 1 of 3 cohorts.

COHORT I: Patients receive cirtuvivint orally (PO) once daily (QD) on days 1-5, 8-12, 15-19, and 22-26 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) at screening. In addition, patients undergo blood sample collection and bone marrow aspiration at screening and on study.

COHORT II: Patients receive cirtuvivint PO QD on days 1, 4, 8, 11, 15, 18, 22, and 25 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA at screening. In addition, patients undergo blood sample collection and bone marrow aspiration at screening and on study.

COHORT III: Patients receive cirtuvivint PO QD on days 1, 4, 8, 11, 15, 18, 22, and 25 and ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA at screening. In addition, patients undergo blood sample collection and bone marrow aspiration at screening and on study.

After completion of study treatment, patients are followed up for 30 days, every 3 months for 2 years then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* In Cohorts I and II, patients must have R/R AML or MDS (venetoclax naïve or venetoclax exposed)

  * Relapsed AML is defined as the appearance of 5% or greater myeloblasts in the bone marrow or peripheral blood after achieving a complete remission (CR), CR with partial hematologic recovery (CRh), or CR with incomplete hematologic recovery (CRi). Patients with a mutation in FLT3, IDH1 or IDH2 must have failed or been intolerant of a corresponding Food and Drug Administration (FDA) approved FLT3, IDH1 or IDH2 inhibitor before enrolling on study. The initial diagnosis of AML is defined by the ELN 2022 criteria, and therefore patients with either AML (peripheral blood or bone marrow blasts ≥ 20% or blasts ≥ 10% with recurrent genetic abnormalities) or MDS/AML (peripheral blood or bone marrow blasts 10-19%) are eligible
  * Refractory AML is defined as failure to achieve a CR, CRh, or CRi after one of the following regimens: (i) 2 cycles of intensive induction chemotherapy with a cytarabine containing regimen (e.g., 7+3, mitoxantrone, etoposide, cytarabine [MEC], high-dose cytarabine [HIDAC], reinduction chemotherapy such as 5 + 2, etc.) or, (ii) 2 cycles of hypomethylating agent (HMA)/venetoclax or low-dose cytarabine (LDAC)/glasdegib or, (iii) ≥ 4 cycles of HMA monotherapy. The initial diagnosis of AML is defined by the ELN 2022 criteria, and therefore patients with either AML (peripheral blood or bone marrow blasts ≥ 20% or blasts ≥ 10% with recurrent genetic abnormalities) or MDS/AML (peripheral blood or bone marrow blasts 10-19%) are eligible
  * Patients with MDS/AML (blasts 10-19%) who progress to AML (blasts ≥ 20%) after treatment will be considered relapsed or refractory MDS/AML, and not as newly-diagnosed AML (i.e. the patients' treatment history for eligibility purposes does not reset)
  * Relapsed MDS is defined as: (i) Intermediate, high, or very high-risk disease by International Prognostic Scoring System-Revised (IPSS-R) and, (ii) Any relapse after achieving any 2023 IWG MDS defined response
  * Refractory MDS is defined as: (i) Intermediate, high, or very high-risk disease by IPSS-R and > 5% blasts in the bone marrow or peripheral blood, (ii) Failure to achieve a response (as per IWG 2006 criteria) after ≥ 4 cycles of HMA monotherapy, or (iii) ≥ 2 cycles of HMA + venetoclax
* In Cohort III, patients must have prior untreated high-risk MDS

  * MDS with > 5% blasts in the bone marrow or peripheral blood AND
  * IPSS-R high or very high-risk disease OR
  * Molecular International Prognostic Scoring System (IPSS-M) high or very high-risk disease
  * No more than one single prior cycle of DNMTi therapy
  * Prior use of erythropoiesis stimulating agents (ESA), thrombopoietin agonists, lenalidomide, and luspatercept are allowed
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of SM08502 (cirtuvivint) in combination with ASTX727 in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3
* Total bilirubin ≤ 2 x institutional upper limit of normal (ULN) (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin; in that case a cut off of ≤ 4 × institutional ULN will be used)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN (unless considered due to organ involvement by the patient's myeloid malignancy; in that case a cut off of ≤ 5 x institutional ULN will be used)
* Glomerular filtration rate (GFR) ≥ 45 mL/min/1.73m^2
* If female, patient must be either:

  * Postmenopausal (surgically sterile or age > 55 years with no menses for 12 or more months without an alternative medical cause or age equal to 55 or less with no menses for 12 or more months without an alternative medical cause and a follicle stimulating hormone [FSH] level > 40 IU/L); or
  * Of children bearing potential. These patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Patient must agree to have a negative urine or serum beta-human chorionic gonadotropin (HCG) test result during screening and repeated within 7 days prior to study drug (local labs are allowed) to be eligible
* The effects of SM08502 (cirtuvivint) and ASTX727 on the developing human fetus are unknown. For this reason, and because these agents are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and during the treatment therapy. Women of childbearing age should agree to use adequate contraception for 7 months after completion of SM08502 (cirtuvivint) administration. For ASTX727, adequate contraception must continue for at least 6 months after last dose of ASTX727. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of the study and at least 4 months after the last dose of SM08502 (cirtuvivint) and 3 months after last dose of ASTX727. Women who are lactating must refrain from breastfeed during the study and at least for two weeks after last dose of ASTX727
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia or abnormal blood counts
* Patients who are receiving any other investigational agents
* Systemic anti-leukemic or other antineoplastic therapy within 14 days of first day of study treatment. If on venetoclax, then a wash-out period of at least five times the half-life of venetoclax is required. Exceptions: No wash-out required for intrathecal chemotherapy, hydroxyurea, cytarabine (Ara-C), or palliative radiation therapy to painful sites of leukemic disease. Patients are not allowed to receive concurrent therapy such as cytotoxic chemotherapy or radiation therapy for another cancer. Patients on hormonal adjuvant therapy for non-metastatic breast and prostate cancer or other minimally-myelosuppressive maintenance therapies for non-metastatic cancer may be eligible at the discretion of the study principal investigator (PI)
* Patient is receiving known inhibitors or activators of flavin-containing monooxygenases (FMO1 or FMO3), and these cannot be stopped at least 5 days prior to SM08502 (cirtuvivint) treatment start. Known inhibitors of FOMO are chlorpromazine and imipramine
* Patient is receiving strong inhibitors or strong inducers of CYP3A4/5 and these cannot be stopped at least 5 days prior to SM08502 (cirtuvivint) treatment start

  * Strong inhibitors include grapefruit juice or grapefruit/grapefruit related citrus fruits (e.g., Seville oranges, pomelos), ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir, nefazodone, lopinavir, troleandomycin, mibefradil, and conivaptan. Examples may be found at the FDA website. Refer to the prescribing information of concomitant medications if in doubt or consult the sponsor for guidance
  * Strong inducers include phenobarbital, rifampin, phenytoin, carbamazepine, rifabutin, rifapentin, clevidipine, and St. John's Wort. Examples may be found at the FDA website. Refer to the prescribing information of concomitant medications if in doubt or consult the sponsor for guidance.
  * While moderate inhibitors or moderate inducers of CYP3A4/5 are not an exclusion criteria for the trial, it is preferred that moderate inhibitors or moderate inducers of CYP3A4/5 be replaced prior to the first dose of SM08502 (cirtuvivint) and during study conduct where this is possible.

    * Moderate inhibitors include erythromycin, ciprofloxacin, verapamil, diltiazem, atazanavir, fluconazole, darunavir, delavirdine, amprenavir, fosamprenavir, aprepitant, imatinib, tofisopam, and cimetidine. Examples may be found at the FDA website. Refer to the prescribing information of concomitant medications if in doubt or consult the sponsor for guidance
    * Moderate inducers include bosentan, efavirenz, etravirine, modafinil, and nafcillin. Examples may be found at the FDA website. Refer to the prescribing information of concomitant medications if in doubt or consult the sponsor for guidance
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SM08502 (cirtuvivint) or ASTX727
* Chronic, active hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: patients with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface [HBs] antigen negative, anti-HBs antibody positive and anti-hepatitis B core [HBc] antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate. Patients who had prior HCV that has been definitively treated with negative HCV viral load prior to study initiation and no evidence of cirrhosis, are allowed to participate. If there is no known history of HBV infection no HBV studies need to be obtained. If there is no known history of HCV infection, no HCV studies need to be obtained
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant and lactating women are excluded from this study because SM08502 (cirtuvivint) is a small molecule inhibitor of CLK DYRK with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SM08502 (cirtuvivint), breastfeeding should be discontinued if the mother is treated with SM08502 (cirtuvivint). These potential risks may also apply to other agents used in this study
* Patients with acute promyelocytic leukemia
* Subject has symptomatic central nervous system (CNS) involvement with AML
* Patient has immediate life-threatening, severe complications of their myeloid malignancy such as uncontrolled bleeding and/or uncontrolled infection
* Patient has significant active cardiac disease within 6 months prior to the start of study treatment, including uncontrolled New York Heart Association (NYHA) class III or IV congestive heart failure; acute coronary syndrome (ACS); and/or stroke
* Left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan obtained within 30 days prior to the start of study treatment
* Patient is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally. Patient needs to be able to swallow pills
* Patient has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
* Subject has prolonged corrected QC (QTc) interval (Fridericia's correction [QTcF]) ≥ 480 ms or known family history of long QT interval syndrome at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to day 28
  The MTD of cirtuvivint as monotherapy in relapsed/refractory (R/R) acute myeloid leukemia (AML) and R/R myelodysplastic syndrome (MDS) (Cohort I and II) and in combination with ASTX727 in frontline MDS (Cohort III). MTD will be defined as the highest dose level at which 0/6 or 1/6 subjects experience a dose-limiting toxicity.
Recommended phase 2 dose (RP2D) | Up to 3 years
  The RP2D will be based on the MTD in both Cohort I and II as well as pharmacokinetic, pharmacodynamic and response data from Cohort I and II.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  AEs will be graded using Common Terminology Criteria for Adverse Events version 5.0 and described by frequency, duration, and severity of treatment-emergent, treatment-related, and serious AEs. All reported toxicities, regardless of attribution, will be summarized by toxicity type and maximum grade, and sorted by number of patients experiencing the toxicity for each dosing cohort and overall.
Clinical response | Up to 5 years after end of treatment
  Clinical response will be assessed based on the 2022 European LeukemiaNet criteria for AML and the 2023 International Working Group criteria for MDS. Clinical response will be described using descriptive statistics. Point estimates and exact binomial 95% confidence intervals (CIs) will be provided for binary endpoints such as response rate in participants treated at MTD.
Event-free survival (EFS) | Up to 1 year
  The Kaplan-Meier method will be used to estimated EFS with its 95% CI.
Overall survival (OS) | Up to 1 year
  The Kaplan-Meier method will be used to estimated OS with its 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Evan C Chen, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (7):
- United States (7):
  - Yale University, New Haven, Connecticut
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm